CLINICAL TRIAL: NCT02715804
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) in Combination With Nab-Paclitaxel Plus Gemcitabine Compared With Placebo Plus Nab-Paclitaxel and Gemcitabine in Subjects With Hyaluronan-High Stage IV Previously Untreated Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of PEGylated Recombinant Human Hyaluronidase in Combination With Nab-Paclitaxel Plus Gemcitabine Compared With Placebo Plus Nab-Paclitaxel and Gemcitabine in Participants With Hyaluronan-High Stage IV Previously Untreated Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HALO-109-301; 2015-004068-13 (EudraCT Number)
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Pancreatic Ductal Carcinoma
Keywords: Pancreatic ductal adenocarcinoma (PDA); Pancreatic ductal carcinoma; PEGylated Recombinant Human Hyaluronidase (PEGPH20); Nab-paclitaxel; Gemcitabine; Metastatic; Stage IV
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Neoplasm Metastasis | interventions — PEGPH20; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PAG: PEGPH20 + nab-Paclitaxel + Gemcitabine (Experimental): Participants will receive 3.0 micrograms/kilogram (μg/kg) PEGPH20 as an intravenous (IV) infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisting of 4 weeks [Week 4 of every cycle will be a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 milligrams/square meter (mg/m^2) nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment will continue until disease progression, unacceptable toxicity, death, or withdrawal of consent.
  Interventions: Other: Biological: PEGylated Recombinant Human Hyaluronidase (PEGPH20); Drug: nab-Paclitaxel; Drug: Gemcitabine
- AG: Placebo + nab-Paclitaxel + Gemcitabine (Placebo Comparator): Participants will receive placebo matching to PEGPH20 as an IV infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisting of 4 weeks [Week 4 of every cycle will be a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 mg/m^2 nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment will continue until disease progression, unacceptable toxicity, death, or withdrawal of consent.
  Interventions: Drug: Placebo; Drug: nab-Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Other: Biological: PEGylated Recombinant Human Hyaluronidase (PEGPH20) — PEGPH20 will be administered as per the dose and schedule specified in the respective arms.
  Arms: PAG: PEGPH20 + nab-Paclitaxel + Gemcitabine
Drug: Placebo — Matching placebo for PEGPH20
  Arms: AG: Placebo + nab-Paclitaxel + Gemcitabine
Drug: nab-Paclitaxel — Nab-paclitaxel will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Abraxane®
Drug: Gemcitabine — Gemcitabine will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Gemzar®

SUMMARY:
The purpose of this study is to compare the efficacy and safety of PEGylated Recombinant Human Hyaluronidase (PEGPH20) combined with nab-paclitaxel plus gemcitabine (PAG treatment), compared with placebo combined with nab-paclitaxel plus gemcitabine (AG treatment), in participants with hyaluronan (HA)-high Stage IV previously untreated pancreatic ductal adenocarcinoma (PDA).

DETAILED DESCRIPTION:
Participants will be randomized in a 2:1 ratio to PAG or AG treatment.

ELIGIBILITY:
Inclusion criteria:

Participants must satisfy all the following inclusion criteria to be enrolled in the study:

1. Signed, written Institutional Review Board/Ethics Committee-approved Informed Consent Form (ICF).
2. Stage IV PDA with histological or cytological confirmation of PDA.
3. Participants must be determined to be HA-high based on archived or fresh tumor core biopsy or sample obtained after the participant has documented metastatic disease. Biopsies/samples must meet the following requirements:

   1. Pancreas tumor biopsies/samples obtained on or after the date that metastatic disease is documented or tumor biopsies/samples from a metastatic lesion are acceptable.
   2. Tumor biopsies or samples must meet the requirements provided in the Study Laboratory Manual with regard to tumor tissue architecture. Note: cytology samples from fine needle aspirates without maintained tissue architecture or brushing biopsies are not acceptable.
   3. Tumor tissue (formalin-fixed paraffin-embedded [FFPE] block preferred) must include enough tumor to make a minimum of 5-10 unstained, consecutive FFPE slides (10 slides are preferred) of 1 archival block that meet specific tissue sample requirements.
4. Radiographic confirmation of Stage IV PDA with at least 1 tumor metastasis measurable on computed tomography (CT) scan or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria, excluding the primary pancreatic lesion.
5. If a participant has had adjuvant/neoadjuvant therapy and/or therapy for locally advanced disease (chemotherapy for non-metastatic pancreatic cancer in combination with or without radiation therapy), tumor recurrence or disease progression must have occurred no sooner than 6 months after completing the last dose of the aforementioned therapies, provided all toxicities have returned to baseline or less than or equal to (≤) Grade 1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Life expectancy greater than or equal to (≥) 3 months.
8. Age ≥18 years.
9. A negative urine or serum pregnancy test within 7 days before Cycle 1, Day 1 (C1D1; first dose of study medication) if female participant is of childbearing potential.
10. Screening clinical laboratory values as follows:

    1. Total bilirubin ≤1.5 times upper limit of normal (ULN) (participants with Gilbert syndrome are eligible independent of bilirubin levels).
    2. Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvate transaminase) ≤2.5 times ULN, (if liver metastases are present, then ≤5 times ULN is allowed).
    3. Serum creatinine ≤2.0 milligrams/deciliter (mg/dL) or calculated creatinine clearance ≥40 milliliters/minute (mL/min).
    4. Serum albumin ≥2.5 grams/deciliter (g/dL).
    5. Prothrombin time or international normalized ratio (INR) within normal limits (±15%), unless participant takes warfarin, in which case prothrombin time or INR result must be within therapeutic range.
    6. Partial thromboplastin time (PTT) within normal limits (±15%).
    7. Hemoglobin ≥9 g/dL (transfusion and erythropoietic agents allowed).
    8. Absolute neutrophil count ≥1,500 cells/cubic millimeter (cells/mm^3).
    9. Platelet count ≥100,000/mm^3.
11. For women of childbearing potential (WOCBP) and for men, agreement to use a highly effective contraceptive method from the time of screening throughout the study until 1 month (WOCBP) or 6 months (men) after administration of the last dose of any study medication. Highly effective contraceptive methods consist of prior sterilization, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), oral or injectable contraceptives, barrier methods, and/or true sexual abstinence.

Exclusion criteria:

Participants are ineligible for enrollment if they meet any of the following exclusion criteria:

1. Clinical evidence of deep vein thrombosis (DVT), pulmonary embolism (PE) or other known thromboembolic (TE) event present during the screening period.

   1. Participants with superficial vein thrombosis are eligible.
   2. Participants with visceral/splanchnic vein thrombosis are still eligible if, in the opinion of the Investigator, the visceral/splanchnic vein thrombosis is primarily associated with the anatomic location of the underlying disease of metastatic pancreatic cancer (there must be primary or metastatic disease in reasonable proximity to the thrombosis, and the Investigator determines that the thrombosis is due to a local tumor event and not a coagulation issue).
2. Previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease.

   a. Palliative radiotherapy for pain control of metastatic bone lesions is allowed.
3. Known central nervous system involvement or brain metastases.
4. New York Heart Association Class III or IV cardiac disease or myocardial infarction within the past 12 months.
5. History of cerebrovascular accident or transient ischemic attack.
6. Clinically significant pre-existing carotid artery disease.
7. Known infection with human immunodeficiency virus, or active infection with hepatitis B or hepatitis C within the past 12 months.
8. Known allergy to hyaluronidase.
9. Current use of megestrol acetate or megestrol acetate-containing drugs (use within 10 days of Day 1).
10. Contraindication to heparin as per institutional guidelines.
11. Women currently pregnant or breastfeeding.
12. Intolerance to dexamethasone.
13. History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ.
14. Any other disease, active, uncontrolled bacterial, viral or fungal infection requiring systemic therapy, metabolic dysfunction, physical examination finding or clinical laboratory finding that leads to reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, or that may affect the interpretation of the results, or that may render the participant at high risk for treatment complications.
15. Immunization with a live vaccine up to 2 weeks prior to Day 1.
16. Hypersensitivity to the active substance or ingredients of PEGPH20, gemcitabine, and nab-paclitaxel.
17. Inability to comply with study and follow-up procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Medical, Regulatory and Drug Safety, Study Director — Halozyme Therapeutics
Locations (217):
- United States (64):
  - University of South Alabama, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - St. Jude Hospital Yorba DBA Linda St. Joseph Heritage Health, Fullerton, California
  - Scripps Clinical Research Services, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - David Geffen School of Medicine (DGSOM) at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - St. Joseph Hospital, Orange, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Pacific Central Coast Health Centers: San Luis Obispo Oncology and Hematology Health Center, San Luis Obispo, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Innovative Clinical Research Institution, Whittier, California
  - Kaiser Permanente Franklin Medical Offices - Denver, Denver, Colorado
  - US Oncology - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - St. Mary's Medical Center, Grand Junction, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Memorial Healthcare System - Memorial Cancer Institute, Hollywood, Florida
  - 21st Century Oncology, Jacksonville, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Fort Wayne Medical Oncology/Hematology, INC., Fort Wayne, Indiana
  - The University Of Kansas Cancer Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Ochsner Health Center, Baton Rouge, Louisiana
  - Ochsner Clinic CCOP, New Orleans, Louisiana
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Joseph's Ambulatory Clinic, Clifton, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - NYU Langone Medical Center - NYU Langone Arena Oncology, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai School of Medicine - The Tisch Cancer Institute, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Rex Cancer Center, Raleigh, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Cancer institute, Pittsburgh, Pennsylvania
  - Baylor College of Medicine - Baylor Clinic, Houston, Texas
  - Scott and White, Temple, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Inova Dwight and Martha Schar Cancer Institute, Fairfax, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Virginia Cancer Institute, Mechanicsville, Virginia
  - Swedish Cancer Institute/ Swedish Health Services, Seattle, Washington
  - University of Washington (UW) - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - University of Wisconsin Health - UW Carbone Cancer Center, Madison, Wisconsin
  - Columbia St. Marys, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Flinders Medical Centre, Bedford, South Australia
  - Bendigo Health Care Group, Bendigo, Victoria
  - Monash Health, Bentleigh East, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
- Belgium (7):
  - Imelda Ziekenhuis, Bonheiden, Antwerpen
  - UZA, Edegem, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Hôpital Erasme, Brussels, Brussels Capital
  - AZ Maria Middelares - Campus Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Un, Liège
- Brazil (11):
  - CENANTRON - Centro Avançado de Tratamento Oncologico, Belo Horizonte, Minas Gerais
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Occ -Oncologia Clínica De Campinas, Campinas, São Paulo
  - Fundação Amaral Cravalho / Hospital Amaral Carvalho, Jaú, São Paulo
  - Fm Abc/ Cepho, Santo André, São Paulo
  - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Fundacao Pio XII Hospital De Câncer de Barretos, Barretos
  - Instituto COI, Rio de Janeiro
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Croatia (2):
  - Klinicki bolnicki centar Zagreb, Zagreb, City of Zagreb
  - Klinicki bolnički centar Sestre milosrdnice, Zagreb
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - FN Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce (Hospital Na Bulovce), Prague
- Odense Universitetshospital, Odense, Region Syddanmark, Denmark
- Estonia (2):
  - East Tallinn Central Hospital Oncology Center, Tallinn, Harju
  - North Estonian Medical Centre Foundation Clinic of Oncology, Tallinn, Harju
- France (15):
  - Centre Eugene Marquis, Rennes, Brittany Region
  - Hospitalier Jean Minjoz, Besançon, Franche-Comté
  - ICM Val d'Aurelle Saint Eloi - Departement Oncologie, Montpellier, Hérault
  - ICO - Site Ren Gauducheau, Saint-Herblain, Loire-Atlantique
  - CHU Estaing, Clermont-Ferrand, Puy-de-Dôme
  - Hopital Edouard Herriot, Lyon, Rhône
  - Institut De Cancerologie Gustave Roussy, Villejuif, Val-de-Marne
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Hôpital Haut-Leveque, Bordeaux
  - Henri Mondor - Albert Chevenier, Créteil
  - Centre Lyon Berard, Lyon
  - Hopital Privé Jean Mermoz, Lyon
  - Institut Mutualiste Montsouris, Paris
  - Pitié Salpetriere Hospital, Paris
  - Hôpital Beaujon, Clichy, Île-de-France Region
- Germany (11):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München - Campus Grosshadern, München, Bavaria
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Uniklinik Köln-Klinik für Gastroenterologie und Hepatologie am Abdominalzentrum, Cologne, North Rhine-Westphalia
  - Universitätsklinik Carl-Gustav-Carus Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Kliniken Essen-Mitte Evang. Huyssens-Stiftung, Essen
  - Universitätsklinikum Halle-Universitätsklinik und Poliklinik, Halle
  - Facharztzentrum Eppendorf, Hamburg
  - Universitätskllinikum Heidelberg, Heidelberg
- Hungary (11):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpo, Szeged, Csongrád megye
  - Petz Aladár Megyei Oktató Kórház, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Egyesített Szent István és Szent László Kórház-Rendelőintéze, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Semmelweis Egyetem - Isz. Bel, Onkológiai Részleg, Budapest
  - Semmelweis Egyetem - Onkohaematológiai Osztály, Budapest
  - Szent Margit Kórház, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Israel (11):
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov, Central District
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva, Central District
  - Hadassah Medical Organisation, Jerusalem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Ha'Emek Medical Center, Afula
  - Soroka Medical Center [Oncology], Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - The Chaim Sheba Medical Center [Oncology], Tel Litwinsky
- Italy (9):
  - U.O. di Oncologia, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas Rozzano, IRCCS, Rozzano, Milano
  - PO di Cremona, ASST di Cremona, Cremona
  - AO S. Martino, IRCCS, IST-Istituto Nazionale Ricerca Sul Cancro, Genova
  - Ieo, Irccs, Milan
  - IRCCS Ospedale S.Raffaele, Milan
  - Istituto Oncologico Veneto IOV-IRCCS, Padua
  - Regina Elena, Istituto Nazionale dei Tumori, IFO, IRCCS, Roma
  - Borgo Roma, Policlinico G.Rossi, AOU Integrata Verona, Verona
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - P.Stradins Clinical University, Riga
  - SIA "Rigas Austrumu Kliniska Universitates Slimnica", Riga
- Lithuania (2):
  - National Cancer Institute, Vilnius, Vilnius County
  - Vilniaus Universiteto ligonines Santariskiu Klinikos, Vilnius, Vilnius County
- Netherlands (4):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Spaarne Gasthuis, Hoofddorp
  - Radboud Universiteit Nijmegen, Nijmegen
- Poland (3):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onko, Brzozów, Podkarpackie Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Warsaw
- South Korea (11):
  - Dong-A University Hospital, Busan, Busan Gwang'yeogsi
  - Keimyung University Dongsan Medical Center, Daegu, Daegu Gwang'yeogsi
  - Seoul National University Bundang Hospital, Seongnam, Gyeonggido
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Gachon University Gil Medical Center, Incheon
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (15):
  - Institut Català d'Oncologia-Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catalá d´Oncología (I.C.O.), L'Hospitalet de Llobregat, Barcelona
  - H.U. de Fuenlabrada, Fuenlabrada, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - H.del Mar, Barcelona
  - H.Sta.Creu i St.Pau, Barcelona
  - H.U.Vall d'Hebrón, Barcelona
  - H.C. S.Carlos, Madrid
  - H.G.U. G. Marañón, Madrid
  - H.U. F. Jiménez Díaz, Madrid
  - H.U. R. y Cajal, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - F.I. Valenciano de Oncología, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - H.U. Miguel Servet, Zaragoza
- Taiwan (5):
  - China Medical University Hospital, Taichung, Taichung Municipality
  - Changhua Christian Hospital, Changhua
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital- Taipei, Taipei
- United Kingdom (15):
  - Addenbrooke's Hospital, Cambridge, Cambridge, Cambridgeshire
  - Peterborough And Stamford Hospitals, Peterborough, Cambridgeshire
  - Beatson West of Scotland Cancer Centre, Glasgow, Glasgow City
  - Sarah Cannon Research Institute UK (SCRI UK), London, London, City of
  - Edinburgh Cancer Centre Western General Hospital, Edinburgh, Midlothian
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Birkenhead, Wirral
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Castle Hill Hospital, Cottingham
  - Coventry Hospital, Coventry
  - Hammersmith Hospital, London
  - The Royal Marsden NHS Foundation - Sutton, London
  - The Royal Marsden NHS Foundation Trust - Chelsea, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - North Wales Cancer Treatment Centre, Rhyl
  - The Christie NHS Foundation Trust, Withington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 492 participants were enrolled from 14 March 2016 through 26 December 2018 in 20 countries.
Pre-assignment Details: A total of 492 participants were enrolled and randomized in 2:1 ratio to received either PAG (PEGPH20 + Nab-paclitaxel + Gemcitabine) or AG (Placebo + Nab-paclitaxel + Gemcitabine).
Groups:
- PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine: Participants received 3.0 micrograms/kilogram (μg/kg) PEGPH20 as an intravenous (IV) infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisted of 4 weeks [Week 4 of every cycle was a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 milligrams/square meter (mg/m^2) nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment was continued until disease progression, unacceptable toxicity, death, or withdrawal of consent (Maximum exposure: 150.1 weeks).
- AG: Placebo + Nab-Paclitaxel + Gemcitabine: Participants received placebo matching to PEGPH20 as an IV infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisting of 4 weeks [Week 4 of every cycle will be a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 mg/m^2 nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment was continued until disease progression, unacceptable toxicity, death, or withdrawal of consent (Maximum exposure: 83.9 weeks).
Period: Overall Study
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Started | 327 | 165
Received at Least 1 Dose of Study Drug | 323 | 158
Safety Population (Received at least 1 dose of study medication, and analyzed according to the treatment they received.) | 325 (3 participants randomized to AG but received PAG) | 156 (1 participant randomized to PAG but received AG)
Completed | 98 | 52
Not Completed | 229 | 113
Not completed — Death | 222 | 106
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Other than specified | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine: Participants received 3.0 μg/kg PEGPH20 as an IV infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisted of 4 weeks [Week 4 of every cycle was a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 mg/m^2 nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment was continued until disease progression, unacceptable toxicity, death, or withdrawal of consent (Maximum exposure: 150.1 weeks).
- Total: Total of all reporting groups
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine | Total
Number analyzed (Participants) | 327 | 165 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.62) | 62.3 (9.50) | 63.3 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 85 | 232
  Male | 180 | 80 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 11 | 35
  Not Hispanic or Latino | 267 | 138 | 405
  Unknown or Not Reported | 36 | 16 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 266 | 126 | 392
  Black or African American | 11 | 5 | 16
  Asian | 33 | 24 | 57
  Other | 17 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause. Overall survival was analyzed using Kaplan-Meier methods.
Time Frame: From randomization until death from any cause (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 327 | 165
months | 11.2 [10.3 to 12.3] | 11.5 [9.0 to 12.5]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization until the first occurrence of radiological disease progression, as determined by the blinded Central Imaging Vendor (CIV) based on Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1, or death from any cause during the treatment period. Disease progression was defined as at least a 20 percent (%) increase in sum of diameters of target lesions, taking as reference the smallest sum on study thus far, nadir (this included baseline sum if that was the smallest on study); Sum must also demonstrate an absolute increase of at least 5 millimeters (mm); Appearance of one or more new lesions; Unequivocal progression of existing non-target lesions. Surviving participants without disease progression were censored for PFS analysis at the date of last evaluable post-baseline tumor assessment. Surviving participants without any post-baseline disease assessment were censored on Day 1. PFS was estimated using Kaplan-Meier method.
Time Frame: From the date of randomization until disease progression or death from any cause (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 327 | 165
months | 7.1 [5.5 to 7.4] | 7.1 [4.8 to 8.3]

3. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response
Description: ORR was defined as percentage of participants who achieved either a complete response (CR) or partial response (PR) as determined by the blinded CIV based on RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until CR or PR (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 327 | 165
percentage of participants | 47.1 [41.6 to 52.7] | 36.4 [29.0 to 44.2]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first objective response of CR or PR until disease progression (as determined by the blinded CIV based on RECIST version 1.1) or death within 14 days of last dose of study treatment or randomization. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study thus far, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions. DOR was analyzed using Kaplan-Meier methods.
Time Frame: From date of first objective response (CR or PR) until date of first disease progression (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 154 | 60
months | 6.1 [5.5 to 7.8] | 7.4 [5.3 to 9.4]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were defined as AEs that begin or worsen in severity during or after the participant's first dose of study treatment and no later than 30 days after the date of the last dose of study treatment and/or any treatment-related AE regardless of the onset date. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From administration of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Population: Safety population included all participants who received at least 1 dose of study medication, and analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 325 | 156
Participants | 325 | 156

6. Secondary Outcome: Number of Participants With Worst Post-Baseline Hematology and Chemistry (Clinical Laboratory Parameters) Severity Grade During the Study
Description: Severity grade associated with a laboratory parameter value was determined using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening. Grade 0 indicates evaluable lab records but not fall into any CTCAE grade for certain CTCAE term. A worst post-baseline grade shift was defined as the worst change that occurred at any measured timepoint during study. Hematology abnormalities: anemia(hemoglobin decreased), lymphocyte count decreased, lymphocyte count increased, neutropenia(neutrophil count decreased), thrombocytopenia(platelet count decreased), and leukopenia(white blood cell decreased). Chemistry abnormalities: hypoalbuminemia, alkaline phosphatase increased, alanine aminotransferase increased, aspartate aminotransferase increased, hyperbilirubinemia, hypo- and hypercalcemia, creatinine increased, hypo- and hyperglycaemia, hypo- and hyperkalemia, hypo- and hypermagnesemia, hypo- and hypernatremia.
Time Frame: as for outcome 5
Population: Safety population included all participants who received at least 1 dose of study medication, and analyzed according to the treatment they actually received. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 325 | 156
Participants
  Anemia: Post-baseline: number analyzed (Participants) | 321 | 155
  Anemia: Post-baseline: Grade 0 | 6 | 3
  Anemia: Post-baseline: Grade 1 | 84 | 41
  Anemia: Post-baseline: Grade 2 | 164 | 74
  Anemia: Post-baseline: Grade 3 | 67 | 37
  Anemia: Post-baseline: Grade 4 | 0 | 0
  Lymphocyte count decreased: Post-baseline: number analyzed (Participants) | 321 | 155
  Lymphocyte count decreased: Post-baseline: Grade 0 | 33 | 17
  Lymphocyte count decreased: Post-baseline: Grade 1 | 83 | 46
  Lymphocyte count decreased: Post-baseline: Grade 2 | 102 | 46
  Lymphocyte count decreased: Post-baseline: Grade 3 | 90 | 40
  Lymphocyte count decreased: Post-baseline: Grade 4 | 13 | 6
  Lymphocyte count increased: Post-baseline: number analyzed (Participants) | 321 | 155
  Lymphocyte count increased: Post-baseline: Grade 0 | 302 | 150
  Lymphocyte count increased: Post-baseline: Grade 1 | 0 | 0
  Lymphocyte count increased: Post-baseline: Grade 2 | 19 | 5
  Lymphocyte count increased: Post-baseline: Grade 3 | 0 | 0
  Lymphocyte count increased: Post-baseline: Grade 4 | 0 | 0
  Neutropenia: Post-baseline: number analyzed (Participants) | 321 | 155
  Neutropenia: Post-baseline: Grade 0 | 85 | 31
  Neutropenia: Post-baseline: Grade 1 | 27 | 11
  Neutropenia: Post-baseline: Grade 2 | 57 | 30
  Neutropenia: Post-baseline: Grade 3 | 98 | 48
  Neutropenia: Post-baseline: Grade 4 | 54 | 35
  Thrombocytopenia: Post-baseline: number analyzed (Participants) | 322 | 155
  Thrombocytopenia: Post-baseline: Grade 0 | 52 | 32
  Thrombocytopenia: Post-baseline: Grade 1 | 134 | 63
  Thrombocytopenia: Post-baseline: Grade 2 | 76 | 36
  Thrombocytopenia: Post-baseline: Grade 3 | 51 | 20
  Thrombocytopenia: Post-baseline: Grade 4 | 9 | 4
  Leukopenia: Post-baseline: number analyzed (Participants) | 321 | 155
  Leukopenia: Post-baseline: Grade 0 | 74 | 32
  Leukopenia: Post-baseline: Grade 1 | 30 | 15
  Leukopenia: Post-baseline: Grade 2 | 100 | 43
  Leukopenia: Post-baseline: Grade 3 | 87 | 51
  Leukopenia: Post-baseline: Grade 4 | 30 | 14
  Hypoalbuminemia (Albumin): Post-baseline: number analyzed (Participants) | 318 | 155
  Hypoalbuminemia (Albumin): Post-baseline: Grade 0 | 19 | 46
  Hypoalbuminemia (Albumin): Post-baseline: Grade 1 | 102 | 62
  Hypoalbuminemia (Albumin): Post-baseline: Grade 2 | 185 | 44
  Hypoalbuminemia (Albumin): Post-baseline: Grade 3 | 12 | 3
  Hypoalbuminemia (Albumin): Post-baseline: Grade 4 | 0 | 0
  Alkaline phosphatase increased: Post-baseline: number analyzed (Participants) | 318 | 155
  Alkaline phosphatase increased: Post-baseline: Grade 0 | 135 | 57
  Alkaline phosphatase increased: Post-baseline: Grade 1 | 114 | 62
  Alkaline phosphatase increased: Post-baseline: Grade 2 | 50 | 26
  Alkaline phosphatase increased: Post-baseline: Grade 3 | 19 | 10
  Alkaline phosphatase increased: Post-baseline: Grade 4 | 0 | 0
  Alanine aminotransferase increased: Post-baseline: number analyzed (Participants) | 318 | 155
  Alanine aminotransferase increased: Post-baseline: Grade 0 | 69 | 33
  Alanine aminotransferase increased: Post-baseline: Grade 1 | 155 | 72
  Alanine aminotransferase increased: Post-baseline: Grade 2 | 43 | 32
  Alanine aminotransferase increased: Post-baseline: Grade 3 | 51 | 17
  Alanine aminotransferase increased: Post-baseline: Grade 4 | 0 | 1
  Aspartate aminotransferase increased:Post-baseline: number analyzed (Participants) | 319 | 155
  Aspartate aminotransferase increased:Post-baseline: Grade 0 | 77 | 28
  Aspartate aminotransferase increased:Post-baseline: Grade 1 | 168 | 96
  Aspartate aminotransferase increased:Post-baseline: Grade 2 | 49 | 17
  Aspartate aminotransferase increased:Post-baseline: Grade 3 | 25 | 13
  Aspartate aminotransferase increased:Post-baseline: Grade 4 | 0 | 1
  Hyperbilirubinemia: Post-baseline: number analyzed (Participants) | 319 | 155
  Hyperbilirubinemia: Post-baseline: Grade 0 | 237 | 125
  Hyperbilirubinemia: Post-baseline: Grade 1 | 36 | 9
  Hyperbilirubinemia: Post-baseline: Grade 2 | 31 | 15
  Hyperbilirubinemia: Post-baseline: Grade 3 | 12 | 6
  Hyperbilirubinemia: Post-baseline: Grade 4 | 3 | 0
  Hypocalcemia (calcium): Post-baseline: number analyzed (Participants) | 318 | 155
  Hypocalcemia (calcium): Post-baseline: Grade 0 | 224 | 119
  Hypocalcemia (calcium): Post-baseline: Grade 1 | 68 | 30
  Hypocalcemia (calcium): Post-baseline: Grade 2 | 22 | 6
  Hypocalcemia (calcium): Post-baseline: Grade 3 | 4 | 0
  Hypocalcemia (calcium): Post-baseline: Grade 4 | 0 | 0
  Hypercalcemia (calcium): Post-baseline: number analyzed (Participants) | 318 | 155
  Hypercalcemia (calcium): Post-baseline: Grade 0 | 278 | 148
  Hypercalcemia (calcium): Post-baseline: Grade 1 | 34 | 6
  Hypercalcemia (calcium): Post-baseline: Grade 2 | 3 | 0
  Hypercalcemia (calcium): Post-baseline: Grade 3 | 3 | 1
  Hypercalcemia (calcium): Post-baseline: Grade 4 | 0 | 0
  Creatinine increased: Post-baseline: number analyzed (Participants) | 318 | 155
  Creatinine increased: Post-baseline: Grade 0 | 267 | 135
  Creatinine increased: Post-baseline: Grade 1 | 45 | 16
  Creatinine increased: Post-baseline: Grade 2 | 6 | 4
  Creatinine increased: Post-baseline: Grade 3 | 0 | 0
  Creatinine increased: Post-baseline: Grade 4 | 0 | 0
  Hypoglycemia (glucose): Post-baseline: number analyzed (Participants) | 320 | 155
  Hypoglycemia (glucose): Post-baseline: Grade 0 | 292 | 140
  Hypoglycemia (glucose): Post-baseline: Grade 1 | 17 | 9
  Hypoglycemia (glucose): Post-baseline: Grade 2 | 7 | 1
  Hypoglycemia (glucose): Post-baseline: Grade 3 | 3 | 1
  Hypoglycemia (glucose): Post-baseline: Grade 4 | 1 | 4
  Hyperglycemia (glucose): Post-baseline: number analyzed (Participants) | 320 | 155
  Hyperglycemia (glucose): Post-baseline: Grade 0 | 31 | 24
  Hyperglycemia (glucose): Post-baseline: Grade 1 | 90 | 45
  Hyperglycemia (glucose): Post-baseline: Grade 2 | 119 | 44
  Hyperglycemia (glucose): Post-baseline: Grade 3 | 76 | 40
  Hyperglycemia (glucose): Post-baseline: Grade 4 | 4 | 2
  Hypokalemia (potassium): Post-baseline: number analyzed (Participants) | 319 | 155
  Hypokalemia (potassium): Post-baseline: Grade 0 | 202 | 104
  Hypokalemia (potassium): Post-baseline: Grade 1 | 89 | 38
  Hypokalemia (potassium): Post-baseline: Grade 2 | 0 | 0
  Hypokalemia (potassium): Post-baseline: Grade 3 | 24 | 11
  Hypokalemia (potassium): Post-baseline: Grade 4 | 4 | 2
  Hyperkalemia (potassium): Post-baseline: number analyzed (Participants) | 319 | 155
  Hyperkalemia (potassium): Post-baseline: Grade 0 | 245 | 122
  Hyperkalemia (potassium): Post-baseline: Grade 1 | 44 | 19
  Hyperkalemia (potassium): Post-baseline: Grade 2 | 21 | 11
  Hyperkalemia (potassium): Post-baseline: Grade 3 | 7 | 3
  Hyperkalemia (potassium): Post-baseline: Grade 4 | 2 | 0
  Hypomagnesemia (magnesium): Post-baseline: number analyzed (Participants) | 318 | 154
  Hypomagnesemia (magnesium): Post-baseline: Grade 0 | 209 | 113
  Hypomagnesemia (magnesium): Post-baseline: Grade 1 | 95 | 36
  Hypomagnesemia (magnesium): Post-baseline: Grade 2 | 9 | 5
  Hypomagnesemia (magnesium): Post-baseline: Grade 3 | 4 | 0
  Hypomagnesemia (magnesium): Post-baseline: Grade 4 | 1 | 0
  Hypermagnesemia (magnesium): Post-baseline: number analyzed (Participants) | 318 | 154
  Hypermagnesemia (magnesium): Post-baseline: Grade 0 | 306 | 150
  Hypermagnesemia (magnesium): Post-baseline: Grade 1 | 8 | 4
  Hypermagnesemia (magnesium): Post-baseline: Grade 2 | 0 | 0
  Hypermagnesemia (magnesium): Post-baseline: Grade 3 | 4 | 0
  Hypermagnesemia (magnesium): Post-baseline: Grade 4 | 0 | 0
  Hyponatremia (sodium): Post-baseline: number analyzed (Participants) | 318 | 155
  Hyponatremia (sodium): Post-baseline: Grade 0 | 96 | 49
  Hyponatremia (sodium): Post-baseline: Grade 1 | 167 | 85
  Hyponatremia (sodium): Post-baseline: Grade 2 | 0 | 0
  Hyponatremia (sodium): Post-baseline: Grade 3 | 54 | 21
  Hyponatremia (sodium): Post-baseline: Grade 4 | 1 | 0
  Hypernatremia (sodium): Post-baseline: number analyzed (Participants) | 318 | 155
  Hypernatremia (sodium): Post-baseline: Grade 0 | 308 | 153
  Hypernatremia (sodium): Post-baseline: Grade 1 | 9 | 2
  Hypernatremia (sodium): Post-baseline: Grade 2 | 0 | 0
  Hypernatremia (sodium): Post-baseline: Grade 3 | 0 | 0
  Hypernatremia (sodium): Post-baseline: Grade 4 | 1 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: ECGs including clinical significance was evaluated by the Investigator. Criteria for clinical significance were as per investigator's discretion.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 325 | 156
Participants | 8 | 4

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included measurement of blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), heart rate, and body weight. Criteria for clinical significance abnormalities were: Heart rate: <50 beats per minute (bpm), >120 bpm, >=30 bpm increase from baseline, >=30 bpm decrease from baseline. SBP: >140 millimeters of mercury (mmHg) and increase from baseline >20 mmHg, >180 mmHg, <90 mmHg and decrease from baseline >10 mmHg. DBP: >90 mmHg and increase from baseline >20 mmHg, >105 mmHg, <60 mmHg and decrease from baseline >10 mmHg. Change in weight: >=5% increase from baseline, >=5% decrease from baseline.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
Number analyzed (Participants) | 325 | 156
Participants
  Heart rate: <50 bpm | 7 | 4
  Heart rate: >120 bpm | 47 | 13
  Heart rate: >=30 bpm increase from baseline | 102 | 26
  Heart rate: >=30 bpm decrease from baseline | 38 | 19
  SBP: >140 mmHg and increase from baseline >20 mmHg | 75 | 37
  SBP: >180 mmHg | 6 | 4
  SBP: <90 mmHg and decrease from baseline >10 mmHg | 60 | 17
  DBP: >90 mmHg and increase from baseline >20 mmHg | 21 | 10
  DBP: >105 mmHg | 8 | 6
  DBP: <60 mmHg and decrease from baseline >10 mmHg | 142 | 56
  Change in weight: >=5% increase from baseline | 85 | 52
  Change in weight: >=5% decrease from baseline | 151 | 57

ADVERSE EVENTS:
Time Frame: From administration of first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 150.1 weeks for PAG, and 83.9 weeks for AG)
Description: Safety population included all participants who received at least 1 dose of study medication, and analyzed according to the treatment they actually received. 3 participants randomized to AG but received PAG, hence included in PAG arm for safety assessment and 1 participant randomized to PAG but received AG, hence included in AG arm for safety assessment.
Groups:
- AG: Placebo + Nab-Paclitaxel + Gemcitabine: Participants received placebo matching to PEGPH20 as an IV infusion, twice weekly for Weeks 1 to 3 of Cycle 1 (each cycle consisting of 4 weeks [Week 4 of every cycle will be a rest week with no treatment]), then once weekly for Weeks 1 to 3 of Cycle 2 and beyond in combination with 125 mg/m^2 nab-paclitaxel as an IV infusion and 1000 mg/m^2 gemcitabine as an IV infusion, once weekly for Weeks 1 to 3 of all treatment cycles. Treatment was continue until disease progression, unacceptable toxicity, death, or withdrawal of consent (Maximum exposure: 83.9 weeks).
Arm/Group | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine | AG: Placebo + Nab-Paclitaxel + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 222/325 | 106/156
Serious Adverse Events (participants affected / at risk) | 187/325 | 80/156
Other Adverse Events (participants affected / at risk) | 198/325 | 73/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine (N=325) | AG: Placebo + Nab-Paclitaxel + Gemcitabine (N=156)
Diarrhoea (Gastrointestinal disorders) | 13 | 7
Abdominal pain (Gastrointestinal disorders) | 10 | 6
Vomiting (Gastrointestinal disorders) | 9 | 5
Colitis (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Ascites (Gastrointestinal disorders) | 4 | 0
Ileus (Gastrointestinal disorders) | 3 | 1
Diverticular perforation (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Jejunal ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 22 | 4
Pneumonia (Infections and infestations) | 10 | 6
Liver abscess (Infections and infestations) | 8 | 2
Septic shock (Infections and infestations) | 6 | 1
Bacteraemia (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 4 | 1
Device related infection (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 2 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 2
Abdominal abscess (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Proteus infection (Infections and infestations) | 1 | 0
Pseudomonas bronchitis (Infections and infestations) | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 10
Anaemia (Blood and lymphatic system disorders) | 9 | 3
Neutropenia (Blood and lymphatic system disorders) | 8 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 23 | 8
Asthenia (General disorders) | 6 | 2
Fatigue (General disorders) | 6 | 1
General physical health deterioration (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 3 | 0
Chills (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 8 | 6
Bile duct obstruction (Hepatobiliary disorders) | 6 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 2
Bile duct stenosis (Hepatobiliary disorders) | 2 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 8 | 3
Hypotension (Vascular disorders) | 4 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 1
Thrombophlebitis superficial (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Vitamin K decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 4 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 2 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0/147 | 1/85 — This is a gender-specific AE. Only female participants were at risk.
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PAG: PEGPH20 + Nab-Paclitaxel + Gemcitabine (N=325) | AG: Placebo + Nab-Paclitaxel + Gemcitabine (N=156)
Oedema peripheral (General disorders) | 198 | 52
Fatigue (General disorders) | 162 | 70
Pyrexia (General disorders) | 94 | 49
Asthenia (General disorders) | 74 | 36
Chills (General disorders) | 25 | 10
Mucosal inflammation (General disorders) | 23 | 7
Peripheral swelling (General disorders) | 7 | 9
Nausea (Gastrointestinal disorders) | 149 | 68
Diarrhoea (Gastrointestinal disorders) | 148 | 73
Vomiting (Gastrointestinal disorders) | 100 | 38
Constipation (Gastrointestinal disorders) | 85 | 58
Abdominal pain (Gastrointestinal disorders) | 80 | 43
Stomatitis (Gastrointestinal disorders) | 34 | 9
Abdominal pain upper (Gastrointestinal disorders) | 23 | 11
Dry mouth (Gastrointestinal disorders) | 22 | 9
Dyspepsia (Gastrointestinal disorders) | 22 | 10
Abdominal distension (Gastrointestinal disorders) | 19 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 166 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 92 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 8
Anaemia (Blood and lymphatic system disorders) | 139 | 70
Neutropenia (Blood and lymphatic system disorders) | 106 | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 90 | 32
Leukopenia (Blood and lymphatic system disorders) | 28 | 15
Decreased appetite (Metabolism and nutrition disorders) | 106 | 42
Hypokalaemia (Metabolism and nutrition disorders) | 51 | 23
Hypoalbuminaemia (Metabolism and nutrition disorders) | 48 | 11
Dehydration (Metabolism and nutrition disorders) | 37 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 37 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 30 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 22 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 10
Neuropathy peripheral (Nervous system disorders) | 64 | 24
Dysgeusia (Nervous system disorders) | 53 | 25
Dizziness (Nervous system disorders) | 46 | 24
Peripheral sensory neuropathy (Nervous system disorders) | 42 | 27
Headache (Nervous system disorders) | 33 | 20
Paraesthesia (Nervous system disorders) | 25 | 17
Platelet count decreased (Investigations) | 73 | 36
Weight decreased (Investigations) | 57 | 14
Neutrophil count decreased (Investigations) | 55 | 39
Alanine aminotransferase increased (Investigations) | 51 | 25
White blood cell count decreased (Investigations) | 44 | 23
Aspartate aminotransferase increased (Investigations) | 34 | 17
Blood alkaline phosphatase increased (Investigations) | 16 | 8
Blood bilirubin increased (Investigations) | 13 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 110 | 59
Rash (Skin and subcutaneous tissue disorders) | 28 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 10
Erythema (Skin and subcutaneous tissue disorders) | 14 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 48 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Urinary tract infection (Infections and infestations) | 28 | 11
Upper respiratory tract infection (Infections and infestations) | 18 | 11
Insomnia (Psychiatric disorders) | 61 | 17
Depression (Psychiatric disorders) | 22 | 11
Anxiety (Psychiatric disorders) | 20 | 11
Hypotension (Vascular disorders) | 46 | 20
Hypertension (Vascular disorders) | 23 | 12
Fall (Injury, poisoning and procedural complications) | 19 | 4

LIMITATIONS AND CAVEATS:
Due to the negative study outcome, development of PEGPH20 was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02715804/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT02715804/SAP_001.pdf